CLINICAL TRIAL: NCT02758080
Title: Pragmatic Clinical Trial of Matching Malignant Hematologic Cancer Patients With Adequate Early Phase Clinical Trials by Next-generation Sequencing
Brief Title: Matching Patients With Hematologic Malignancy to Adequate Clinical Trials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: The Korea Health Technology R&D Project through the Korea Health Industry Development Institute (Unknown); Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Youngil Koh, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1690
Record Dates: First submitted 2016-04-15; First posted 2016-05-02 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Hematologic Malignancies
Keywords: Personalized medicine; Next generation sequencing
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matched (Experimental): A molecular profile is identified using next generation sequencing. A participant in this arm is assigned to early clinical trial studying targeted agent, which is anticipated to have the best response rate.
  Interventions: Other: Matching on the basis of molecular analysis
- Not matched (Other): A participants in this arm is assigned to a clinical trial at physician's choice.
  Interventions: Other: Matching on the basis of physician's choice

INTERVENTIONS:
Other: Matching on the basis of molecular analysis
  Arms: Matched
Other: Matching on the basis of physician's choice
  Arms: Not matched

SUMMARY:
A molecular profile of a patient with hematologic malignancy, for whom standard-of-care had failed, is identified using next generation sequencing. Patients are assigned to early clinical trials of targeted agent based on the molecular profiling or physician's choice. The improvement of outcomes in the intention-to-treat population is investigated.

DETAILED DESCRIPTION:
Most of hematologic malignancy patient becomes incurable with standard treatment during their disease course. Although these patients are recommended to participate in an early phase clinical trials, the response rate have reported be only 4 to 6 percent. Over several decades, a lot of cancer driving mutations has been identified, and targeted agents directed at the mutations are continuously developed and studied in many clinical trials. Most of the clinical trials recruited participants regardless of mutational status of them. Recently, however, participants has been recruited in recent clinical trials according to the presence of specific mutations. The response rate of these recent clinical trials is 12-75%.

In this pragmatic clinical trial, cancer driving mutations in hematologic malignancy patients is identified using next generation sequencing, and assign patients to an appropriate clinical trial which is anticipated to exhibit the best response. The improvement of outcome of this biomarker-driven assignment is investigated.

ELIGIBILITY:
Inclusion Criteria:

* adults with > 18 years old
* incurable hematologic malignancy patients who failed to respond to standard treatment
* patients who agreed to this protocol with informed consent
* Eastern Cooperative Oncology Group performance status ≤ 3
* Tolerable major organ function determined by laboratory examination

Exclusion Criteria:

* Expected survival < 3 months
* patients with poor compliance
* patients who can not give an informed consent
* patients who are participating another clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | one year
  Response evaluation is based on the criteria suggested in a clinical trial to which a participant is assigned.

SECONDARY OUTCOMES:
Types of identified molecular profile | one year
Overall survival | one year
Progression-free survival | one year
Toxicity profile | one year
  according to CTCAE version 4.0
Frequencies of identified molecular profile | one year

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horstmann E, McCabe MS, Grochow L, Yamamoto S, Rubinstein L, Budd T, Shoemaker D, Emanuel EJ, Grady C. Risks and benefits of phase 1 oncology trials, 1991 through 2002. N Engl J Med. 2005 Mar 3;352(9):895-904. doi: 10.1056/NEJMsa042220. PMID 15745980
- [Background] Kola I, Landis J. Can the pharmaceutical industry reduce attrition rates? Nat Rev Drug Discov. 2004 Aug;3(8):711-5. doi: 10.1038/nrd1470. No abstract available. PMID 15286737
- [Background] Reichert JM, Wenger JB. Development trends for new cancer therapeutics and vaccines. Drug Discov Today. 2008 Jan;13(1-2):30-7. doi: 10.1016/j.drudis.2007.09.003. Epub 2007 Oct 18. PMID 18190861
- [Background] Tsimberidou AM, Iskander NG, Hong DS, Wheler JJ, Falchook GS, Fu S, Piha-Paul S, Naing A, Janku F, Luthra R, Ye Y, Wen S, Berry D, Kurzrock R. Personalized medicine in a phase I clinical trials program: the MD Anderson Cancer Center initiative. Clin Cancer Res. 2012 Nov 15;18(22):6373-83. doi: 10.1158/1078-0432.CCR-12-1627. Epub 2012 Sep 10. PMID 22966018
- [Background] Tan DS, Thomas GV, Garrett MD, Banerji U, de Bono JS, Kaye SB, Workman P. Biomarker-driven early clinical trials in oncology: a paradigm shift in drug development. Cancer J. 2009 Sep-Oct;15(5):406-20. doi: 10.1097/PPO.0b013e3181bd0445. PMID 19826361
- [Background] Baselga J, Tripathy D, Mendelsohn J, Baughman S, Benz CC, Dantis L, Sklarin NT, Seidman AD, Hudis CA, Moore J, Rosen PP, Twaddell T, Henderson IC, Norton L. Phase II study of weekly intravenous recombinant humanized anti-p185HER2 monoclonal antibody in patients with HER2/neu-overexpressing metastatic breast cancer. J Clin Oncol. 1996 Mar;14(3):737-44. doi: 10.1200/JCO.1996.14.3.737. PMID 8622019
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Flaherty KT, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, O'Dwyer PJ, Lee RJ, Grippo JF, Nolop K, Chapman PB. Inhibition of mutated, activated BRAF in metastatic melanoma. N Engl J Med. 2010 Aug 26;363(9):809-19. doi: 10.1056/NEJMoa1002011. PMID 20818844
- [Background] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- [Background] Krop IE, Beeram M, Modi S, Jones SF, Holden SN, Yu W, Girish S, Tibbitts J, Yi JH, Sliwkowski MX, Jacobson F, Lutzker SG, Burris HA. Phase I study of trastuzumab-DM1, an HER2 antibody-drug conjugate, given every 3 weeks to patients with HER2-positive metastatic breast cancer. J Clin Oncol. 2010 Jun 1;28(16):2698-704. doi: 10.1200/JCO.2009.26.2071. Epub 2010 Apr 26. PMID 20421541
- [Background] Kurzrock R, Sherman SI, Ball DW, Forastiere AA, Cohen RB, Mehra R, Pfister DG, Cohen EE, Janisch L, Nauling F, Hong DS, Ng CS, Ye L, Gagel RF, Frye J, Muller T, Ratain MJ, Salgia R. Activity of XL184 (Cabozantinib), an oral tyrosine kinase inhibitor, in patients with medullary thyroid cancer. J Clin Oncol. 2011 Jul 1;29(19):2660-6. doi: 10.1200/JCO.2010.32.4145. Epub 2011 May 23. PMID 21606412
- [Background] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- [Background] LoRusso PM, Rudin CM, Reddy JC, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Chang I, Darbonne WC, Graham RA, Zerivitz KL, Low JA, Von Hoff DD. Phase I trial of hedgehog pathway inhibitor vismodegib (GDC-0449) in patients with refractory, locally advanced or metastatic solid tumors. Clin Cancer Res. 2011 Apr 15;17(8):2502-11. doi: 10.1158/1078-0432.CCR-10-2745. Epub 2011 Feb 7. PMID 21300762